CLINICAL TRIAL: NCT02698917
Title: Carbon Dioxide, Oxygen and Mean Arterial Pressure After Cardiac Arrest and Resuscitation - Targeting High vs. Low Normal Values
Brief Title: Carbon Dioxide, Oxygen and Mean Arterial Pressure After Cardiac Arrest and Resuscitation
Acronym: COMACARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Laerdal Foundation (Other); The Finnish Medical Association (Other); Orion Research Foundation (Unknown); Finnish Society of Anaesthesiologists (Unknown)
Responsible Party: Principal Investigator, Pekka Jakkula, MD, Helsinki University Central Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 15/2015
Record Dates: First submitted 2016-01-26; First posted 2016-03-04 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Out-of-Hospital Cardiac Arrest
Keywords: Out-of-Hospital Cardiac Arrest; Resuscitation; Hypoxia-Ischemia, Brain
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Hypoxia-Ischemia, Brain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The physician determining neurological outcome at six months after cardiac arrest is blinded to the study group allocations
Oversight: Data Monitoring Committee: No

ARMS (8):
- Group 1 (Active Comparator): Low normal PaCO2, low normal PaO2, low normal MAP
  Interventions: Other: Low normal PaCO2; Other: Low normal PaO2; Other: Low normal MAP
- Group 2 (Active Comparator): High normal PaCO2, low normal PaO2, low normal MAP
  Interventions: Other: High normal PaCO2; Other: Low normal PaO2; Other: Low normal MAP
- Group 3 (Active Comparator): Low normal PaCO2, high normal PaO2, low normal MAP
  Interventions: Other: Low normal PaCO2; Other: High normal PaO2; Other: Low normal MAP
- Group 4 (Active Comparator): High normal PaCO2, high normal PaO2, low normal MAP
  Interventions: Other: High normal PaCO2; Other: High normal PaO2; Other: Low normal MAP
- Group 5 (Active Comparator): Low normal PaCO2, low normal PaO2, high normal MAP
  Interventions: Other: Low normal PaCO2; Other: Low normal PaO2; Other: High normal MAP
- Group 6 (Active Comparator): High normal PaCO2, low normal PaO2, high normal MAP
  Interventions: Other: High normal PaCO2; Other: Low normal PaO2; Other: High normal MAP
- Group 7 (Active Comparator): Low normal PaCO2, high normal PaO2, high normal MAP
  Interventions: Other: Low normal PaCO2; Other: High normal PaO2; Other: High normal MAP
- Group 8 (Active Comparator): High normal PaCO2, high normal PaO2, high normal MAP
  Interventions: Other: High normal PaCO2; Other: High normal PaO2; Other: High normal MAP

INTERVENTIONS:
Other: Low normal PaCO2 — 4.5-4.7 kPa
  Arms: Group 1; Group 3; Group 5; Group 7
Other: High normal PaCO2 — 5.8-6.0 kPa
  Arms: Group 2; Group 4; Group 6; Group 8
Other: Low normal PaO2 — 10-15 kPa
  Arms: Group 1; Group 2; Group 5; Group 6
Other: High normal PaO2 — 20-25 kPa
  Arms: Group 3; Group 4; Group 7; Group 8
Other: Low normal MAP — 65-75 mmHg
  Arms: Group 1; Group 2; Group 3; Group 4
Other: High normal MAP — 80-100 mmHg
  Arms: Group 5; Group 6; Group 7; Group 8

SUMMARY:
The COMACARE trial is a pilot multicenter randomized trial to assess the feasibility and effect on brain injury markers of targeting low or high normal arterial oxygen tension (PaO2), arterial carbon dioxide tension (PaCO2) and mean arterial pressure (MAP) in comatose, mechanically ventilated patients after out-of-hospital cardiac arrest. Using factorial design, participants are randomized at admission to intensive care unit to one of eight groups targeting either low or high normal values of PaO2, PaCO2 and MAP for 36 h. In this way, investigators will be assessing the feasibility and effect of all three variables at the same time.

The primary outcome is serum concentration of neuron-specific enolase (NSE) at 48 h after cardiac arrest. Feasibility outcome is between-group separation in PaO2, PaCO2 and MAP levels. Secondary outcomes include continuous monitoring of cerebral oxygenation, EEG and ECG for 48 h, the levels of NSE, S100B and cardiac troponin at randomization and 24, 48 and 72 h after cardiac arrest and neurological assessment at 6 months after cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Witnessed out-of-hospital cardiac arrest with ventricular fibrillation (VF) or ventricular tachycardia (VT) as the initial rhythm
* Delay of return of spontaneous circulation (ROSC) 10-45 min from the start of the arrest
* Confirmed or suspected cardiac origin
* Mechanical ventilation
* Markedly impaired level of consciousness (no response to verbal commands and Glasgow coma scale [GCS] motor score < 5)
* Deferred consent possible or likely
* Active intensive care initiated, including targeted temperature management (33-36 C)

Exclusion Criteria:

* Probable withdrawal of active ICU care due to terminal illness or poor prognosis because of severely reduced functional status before cardiac arrest
* Confirmed or suspected intracranial pathology and/or suspicion of raised intracranial pressure
* Pregnancy
* Severe oxygenation problem (PaO2 / FiO2 < 100 mmHg)
* Severe COPD

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
Neuron-specific enolase (NSE) serum concentration | 48 hour after cardiac arrest

SECONDARY OUTCOMES:
Neuron-specific enolase (NSE) serum concentration | At randomization and 24 and 72 hour after cardiac arrest
S100B protein serum concentration | At randomization and 24, 48 and 72 hour after cardiac arrest
Cardiac troponin (TnT) serum concentration | At randomization and 24, 48 and 72 hour after cardiac arrest
Cerebral oxygenation monitoring using near infrared spectroscopy (NIRS) monitoring | For 48 hour after admission to ICU
Continuous electroencephalography (EEG) monitoring | For 48 hour after admission to ICU
Functional status using cerebral performance category (CPC) classification | At 30 days and 6 months after cardiac arrest

OTHER OUTCOMES:
Between-group separation in PaCO2 | Every 3 hour for 36 hour after admission to ICU
Between-group separation in PaO2 | Every 3 hour for 36 hour after admission to ICU
Between-group separation in MAP | Every 1 hour for 36 hour after admission to ICU

CONTACTS AND LOCATIONS:
Overall Officials: Matti Reinikainen, Associate Professor, Study Director — Kuopio University Hospital
Locations (7):
- Aarhus University Hospital, Aarhus, Denmark
- Finland (6):
  - Helsinki University Hospital, Helsinki
  - North Karelia Central Hospital, Joensuu
  - Central Finland Central Hospital, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - Päijät-Häme Central Hospital, Lahti
  - Tampere University Hospital, Tampere

REFERENCES:
- [Derived] Laurikkala J, Ameloot K, Reinikainen M, Palmers PJ, De Deyne C, Bert F, Dupont M, Janssens S, Dens J, Hastbacka J, Jakkula P, Loisa P, Birkelund T, Wilkman E, Vaara ST, Skrifvars MB. The effect of higher or lower mean arterial pressure on kidney function after cardiac arrest: a post hoc analysis of the COMACARE and NEUROPROTECT trials. Ann Intensive Care. 2023 Nov 21;13(1):113. doi: 10.1186/s13613-023-01210-0. PMID 37987871
- [Derived] Humaloja J, Lahde M, Ashton NJ, Reinikainen M, Hastbacka J, Jakkula P, Friberg H, Cronberg T, Pettila V, Blennow K, Zetterberg H, Skrifvars MB; COMACARE Study Groups. GFAp and tau protein as predictors of neurological outcome after out-of-hospital cardiac arrest: A post hoc analysis of the COMACARE trial. Resuscitation. 2022 Jan;170:141-149. doi: 10.1016/j.resuscitation.2021.11.033. Epub 2021 Dec 1. PMID 34863908
- [Derived] Laurikkala J, Aneman A, Peng A, Reinikainen M, Pham P, Jakkula P, Hastbacka J, Wilkman E, Loisa P, Toppila J, Birkelund T, Blennow K, Zetterberg H, Skrifvars MB. Association of deranged cerebrovascular reactivity with brain injury following cardiac arrest: a post-hoc analysis of the COMACARE trial. Crit Care. 2021 Sep 28;25(1):350. doi: 10.1186/s13054-021-03764-6. PMID 34583763
- [Derived] Ameloot K, Jakkula P, Hastbacka J, Reinikainen M, Pettila V, Loisa P, Tiainen M, Bendel S, Birkelund T, Belmans A, Palmers PJ, Bogaerts E, Lemmens R, De Deyne C, Ferdinande B, Dupont M, Janssens S, Dens J, Skrifvars MB. Optimum Blood Pressure in Patients With Shock After Acute Myocardial Infarction and Cardiac Arrest. J Am Coll Cardiol. 2020 Aug 18;76(7):812-824. doi: 10.1016/j.jacc.2020.06.043. PMID 32792079
- [Derived] Jakkula P, Hastbacka J, Reinikainen M, Pettila V, Loisa P, Tiainen M, Wilkman E, Bendel S, Birkelund T, Pulkkinen A, Backlund M, Heino S, Karlsson S, Kopponen H, Skrifvars MB. Near-infrared spectroscopy after out-of-hospital cardiac arrest. Crit Care. 2019 May 14;23(1):171. doi: 10.1186/s13054-019-2428-3. PMID 31088512
- [Derived] Jakkula P, Reinikainen M, Hastbacka J, Loisa P, Tiainen M, Pettila V, Toppila J, Lahde M, Backlund M, Okkonen M, Bendel S, Birkelund T, Pulkkinen A, Heinonen J, Tikka T, Skrifvars MB; COMACARE study group. Targeting two different levels of both arterial carbon dioxide and arterial oxygen after cardiac arrest and resuscitation: a randomised pilot trial. Intensive Care Med. 2018 Dec;44(12):2112-2121. doi: 10.1007/s00134-018-5453-9. Epub 2018 Nov 14. PMID 30430209
- [Derived] Jakkula P, Reinikainen M, Hastbacka J, Pettila V, Loisa P, Karlsson S, Laru-Sompa R, Bendel S, Oksanen T, Birkelund T, Tiainen M, Toppila J, Hakkarainen A, Skrifvars MB; COMACARE study group. Targeting low- or high-normal Carbon dioxide, Oxygen, and Mean arterial pressure After Cardiac Arrest and REsuscitation: study protocol for a randomized pilot trial. Trials. 2017 Oct 30;18(1):507. doi: 10.1186/s13063-017-2257-0. PMID 29084585